CLINICAL TRIAL: NCT00999050
Title: Laparoscopic Gastric Bypass for Type 2 Diabetes Mellitus: a Pilot Prospective Study in Overweight and Mildly Obese Subjects
Brief Title: Laparoscopic Gastric Bypass for Type 2 Diabetes Mellitus With Body Mass Index (BMI) < 35
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Francesco Rubino, MD, Assistant Professor, Weill Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0906010450
Record Dates: First submitted 2009-10-14; First posted 2009-10-21 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type two diabetes; gastric bypass surgery; overweight or moderately obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- diabetic pts <35BMI (Experimental): All patients will be in a single arm receiving bypass surgery to assist with diabetes management
  Interventions: Procedure: Gastric bypass for diabetic patients <35 BMI

INTERVENTIONS:
Procedure: Gastric bypass for diabetic patients <35 BMI — The operation is performed under general anesthesia. It is done laparoscopically, meaning that several small openings are made in the abdomen for insertion of long, thin surgical instruments, one with an attached camera. The operation is video monitored. The top of the stomach is divided across, leaving a small pouch for food. The rest of the stomach remains but can receive no food. The gut is divided just past the stomach, and it is attached to the small stomach pouch so that food can get back into the bowel. A second connection is made so that the bile and digestive juices pass into the bowel with the food.
  Other Names: gastric bypass surgery

SUMMARY:
The aim of this study is to evaluate the effect of Roux-en-y gastric bypass (RYGB) in controlling diabetes in subjects with mild obesity (BMI 26-35). The primary endpoint will be the reduction of HbA1c (< 7%), a standard measure of diabetes control; the secondary endpoints will be changes blood sugar , vitamin levels, insulin, c-peptide, and lipids levels, as well as retinal eye examinations, urinalysis to assess kidney function, carotid ultrasound as a marker of cardiovascular function, and alterations in diabetic medications. Fifty subjects with medically documented type 2 Diabetes Mellitus (T2DM) with BMIs between 26 and 35 will undergo standard laparoscopic RYGB. Prior and after surgery, the subjects will undergo a clinical evaluation in regard to the primary and secondary endpoints listed. The pre-surgery evaluation is directed toward establishing the existence of diabetes related complications prior to surgery. After surgery subjects will be closely monitored for complications and required changes in their diabetes management. Repeat assessments will be made at 1, 3, 6, and 12 months and at two years.

DETAILED DESCRIPTION:
The primary endpoint will be the reduction of HbA1c and secondary endpoints will be multiple associated parameters as listed below. A group of 50 subjects with medically documented T2DM and BMI of 26-35 will undergo standard laparoscopic RYGB. Prior to surgery, the subjects will undergo the standard pre-operative work up required for conventional bariatric surgery. This includes full history and physical exam, medical/cardiac clearances as needed, nutrition consultation and a gastrointestinal consultation for upper endoscopy. After thorough explanation an approved informed consent will be signed. Baseline parameters, as listed below, will be measured for each subject to identify possible complications of diabetes prior to the surgical intervention..

After surgery perioperative complications will be monitored and required modifications of diabetes management advised. Followed up measurements at 1, 3, 6, 12, and 24 months is consistent with standard clinical practice guidelines. Data analysis will be ongoing to observe the effects of the surgical intervention on glucose homeostasis.

* Baseline parameters
* History and Physical Exam
* Weight/BMI/ body composition with the Tanita 310.
* Waist Circumference
* Blood Pressure
* CBC
* HbA1c
* Fasting glucose
* Vitamin B6, B12, Folate,and Iron status
* Lipid Profile -total cholesterol, HDL, LDL, triglyceride
* Fasting Insulin and C-peptide
* Stimulated C-peptide
* EKG
* Retinal exam
* Urinalysis (assess for proteinuria and microalbuminuria)
* Comprehensive foot exam
* Medications and dosage
* Quality of Life Score (SF-36)
* Carotid ultrasound (intima-media thickness)

Follow-up:

4 Weeks:

* Physical Examination, wound check, Body weight, BMI,
* Glucose Diary (pre and postprandial glucose levels as required)
* Insulin and C-peptide
* Lipid profile
* Medication use

  3 Months, 6 months,

Same as above plus:

* HbA1c
* Vitamin levels and iron status
* Retinal exam
* Annually the baseline measurements will be repeated

ELIGIBILITY:
Inclusion Criteria:

Adult males and females who meet the following inclusion criteria will be offered the opportunity to participate in the study:

1. Diagnosis of type 2 Diabetes Mellitus (T2DM) confirmed by the following criteria:

   1. normal or high C-peptide level (> 0.9 ng/ml) to exclude type 1 Diabetes Mellitus
   2. positive glucagon test to confirm T2DM
   3. fasting plasma glucose of 126 mg/dl or more on at least two occasions
2. Body mass index (BMI) 26 kg/m2 or greater, and less than 35 kg/m2
3. History of T2DM for not longer than 8 years, as long-standing disease beyond 8 years correlates with failure to achieve diabetes resolution after gastric bypass
4. No contraindication for surgery or general anesthesia as determined by a multidisciplinary bariatric surgery team (surgeon, anesthesiologist, internist, dietitian, psychologist)
5. Between 18 and 65 year of age
6. Able to provide informed consent
7. If a female with reproductive potential, she has to agree to use a reliable method of birth control for at least one year from the date of surgery

Exclusion Criteria

Subjects who meet any of the following exclusion criteria will not be eligible to participate in the study:

1. Enrollment in another clinical study, which involves an investigational drug
2. Diagnosis of type 1 Diabetes Mellitus or other genetic forms of Diabetes Mellitus
3. Significant renal failure of chronic liver disease (except NAFLD)
4. Major psychological disorders
5. Pregnancy - all female subjects will have serum beta-hCG prior to operation, and must use birth control of their choice to avoid pregnancy during the first year after surgery
6. Previous gastric or esophageal surgery
7. Immunosuppressive drugs including corticosteroids
8. Coagulopathy defined as an INR > 1.5 or platelet count < 50,000/µl
9. Anemia defined as a Hb <10.0 g/dl
10. Inflammatory bowel diseases or other medical condition that would serve as a contraindication to gastric bypass (eg. celiac sprue, pancreatic insufficiency)
11. A severe concurrent illness that is likely to limit life or require extensive systemic treatment (e.g. cancer)
12. A pre-existing major complication of diabetes:

    1. unstable, proliferative retinopathy
    2. severe autonomic cardiac neuropathy or intestinal neuropathy
    3. Myocardial infarction within the previous year, current unstable angina, or poorly-controlled congestive heart failure (Stage III)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C changes | Post gastric bypass operation

SECONDARY OUTCOMES:
improvement in glycemic control | 1 to two years

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College New York Prysbyterian Hosptial, New York, New York, United States

REFERENCES:
- [Background] Cohen R, Pinheiro JS, Correa JL, Schiavon CA. Laparoscopic Roux-en-Y gastric bypass for BMI < 35 kg/m(2): a tailored approach. Surg Obes Relat Dis. 2006; 2(3):401-4. Cohen RV, Schiavon CA, Pinheiro JS, Correa JL, Rubino F. Duodenal-jejunal bypass for the treatment of type 2 diabetes in patients with body mass index of 22-34 kg/m2: a report of 2 cases. Surg Obes Relat Dis. 2007; 3(2): 195-7. Lee WJ, Wang W, Lee YC, Huang MT, Ser KH, Chen JC. Effect of laparoscopic mini-gastric bypass for type 2 diabetes mellitus: comparison of BMI>35 and <35 kg/m2. J Gastrointest Surg. 2008; 12(5): 945-52. Scopinaro N, Papadia F, Marinari G, Camerini G, Adami G. Long-term control of type 2 diabetes mellitus and the other major components of the metabolic syndrome after biliopancreatic diversion in patients with BMI < 35 kg/m2. Obes Surg. 2007; 17(2): 185-92. Chiellini C, Rubino F, Castagneto M, Nanni G, Mingrone G. The effect of bilio-pancreatic diversion on type 2 diabetes in patients with BMI <35 kg/m2. Diabetologia. 2009; 52(6): 1027-30.